CLINICAL TRIAL: NCT05404113
Title: Comparison of Sustained Natural Apophyseal Glide and Deep Friction Massage in Patients With Cervicogenic Headache
Brief Title: Sustained Natural Apophyseal Glide and Deep Friction Massage in Patients With Cervicogenic Headache
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/01251 Aroosha Akbar
Record Dates: First submitted 2022-04-21; First posted 2022-06-03 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Headache Disorders
Keywords: Sustained natural apophyseal glide/SNAG; deep friction massage; Cervicogenic headache
MeSH Terms: conditions — Headache Disorders; Post-Traumatic Headache

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sustained natural apophyseal glide (Experimental): Mulligan's C1-C2 self-SNAG + Conventional PT
  Interventions: Other: sustained natural apophyseal glide
- deep friction massage (Experimental): Cyriax deep friction massage+ Conventional PT
  Interventions: Other: deep friction massage

INTERVENTIONS:
Other: sustained natural apophyseal glide — Mulligan's C1-C2 self-SNAG+ strengthening exercises for anterior and posterior neck muscles (extension, flexion, rotation, lateral flexion) Frequency: 2-3 times/week for 3 weeks Intensity: moderate intensity (pain free) Time: 20 minutes/session Type: Mobilization with movement SNAG Conventional PT including strengthening exercises neck muscles 10 repetitions, 1 set Resisted neck flexion, extension, lateral flexion, rotation Frequency: 2-3 times/week for 3 weeks Intensity: moderate-high intensity (depending on pain tolerance) Time: 10 minutes/session Type: Strengthening Exercise
  Arms: sustained natural apophyseal glide
Other: deep friction massage — Cyriax deep friction massage+ strengthening exercises for anterior and posterior neck muscles (extension, flexion, rotation, lateral flexion) Frequency: 2-3 times/week for 3 weeks Intensity: moderate-high intensity (depending on pain tolerance) Time: 20 minutes/session Type: Deep soft tissue massage Conventional PT including strengthening exercises neck muscles 10 repetitions, 1 set Resisted neck flexion, extension, lateral flexion, rotation Frequency: 2-3 times/week for 3 weeks Intensity: moderate-high intensity (depending on pain tolerance) Time: 10 minutes/session Type: Strengthening Exercise
  Arms: deep friction massage

SUMMARY:
The aim of this randomized controlled trial is to compare the effects of sustained natural apophyseal glide and deep friction massage in patients with cervicogenic headache for reducing pain, enhancing cervical range of motion and improving sleep quality.

DETAILED DESCRIPTION:
Cervicogenic headache CGH is defined as the headache which arises from lesion occurring in the upper three cervical vertebrae and its associated soft tissue structures. Sleep disturbance has been continuously associated with headaches. CGH is a secondary type of headache as classified by the International Classification of Headache Disorders IHD. Physical and manual modes of therapy are important therapeutic modalities for the acute rehabilitation of cervicogenic headache.

The "mobilization with movement" concept, known as the Mulligan concept, is entirely distinct from other forms of manual therapy. Mulligan described the sustained natural apophyseal glide (SNAG) on the joint with active movement done by the patient in the direction of the symptoms. This glide should be pain-free, with proper force applied by a trained person). Efficacy of SNAG C1-C2 has been proven in patients experiencing acute to subacute CGH for both short and long-term periods. Mulligan recommended that mobilization should be done towards the restricted site or in the direction of symptom reproduction, which is difficult to find in patients experiencing headache and dizziness in only one direction. There is evidence that mobilizing symptomatic and asymptomatic cervical levels result in immediate improvement of pain and segmental mobility at the same level as well as adjacent areas.

James Cyriax proposed a treatment technique, Deep friction massage which has a significant effect in pain relieving. Cyriax friction massage is a widely known and used technique in the field of chronic pain management. It is a type of connective tissue massage applied to the soft tissue structures such as tendon, muscle bellies, musculotendinous junction, ligaments and joint capsules. This approach targets muscles both superficial and deep that can be contributing to headache. Muscles (such as trapezius, sternocleidomastoid, levator scapulae, and deep neck flexors) that contribute in developing CGH can be targeted using this technique.

Mulligan's SNAG is a sustained glide that includes a sustained facet glide and active movement simultaneously; this technique targets the joint as well as muscle's active contraction. This reinforces the cervical lesion thus reducing CGH. Deep friction massage enables the skin, fascia; muscles to be involved in order to improve circulation thus promote healing. These techniques will help relieve cervicogenic headache and a proper comparison will be made which is novel. The effectiveness of these techniques in relieving headache, improving ROM and sleep quality will be investigated.

ELIGIBILITY:
Inclusion Criteria; Both males & females. Aged 18 years old and above. International Classification of Headache Disorders (ICHD-III) Diagnostic Criteria for cervicogenic headache

Evidence of causation demonstrated by at least two of the following:

* headache has developed in temporal relation to the onset of the cervical disorder or appearance of the lesion
* headache has significantly improved or resolved in parallel with improvement in or resolution of the cervical disorder or lesion
* cervical range of motion is reduced and headache is made significantly worse by provocative maneuvers (Flexion Rotation Test FRT)
* headache is abolished following diagnostic blockade of a cervical structure or its nerve supply • A headache frequency that is more than 2 months.

Exclusion Criteria:

* Bilateral headaches (typifying tension headache) & features suggestive of migraine.
* Known cases of Hydrocephalus.
* Known cases of neurological impairments.
* Known cases of malignancy.
* Involvement in physiotherapy or chiropractic treatment for headache in the previous 12 months.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2022-09-14 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-04-02 (Actual)

PRIMARY OUTCOMES:
Neck Disability Index NDI | 3 weeks
  This questionnaire gives us the information as to how the neck pain has affected one's ability to manage in everyday life. Questions are scored on a vertical scale of 0-5, Likert type scale. A score of 22% or more is considered a significant ADL disability.

SECONDARY OUTCOMES:
Visual Analogue Scale VAS | 3 weeks
  The pain VAS is a unidimensional measure of pain intensity, which has been widely used in diverse adult populations.
  It takes less than a minute to administer. Using a ruler, the score is determined by measuring the distance (mm) on the 10-cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-100. A higher score indicates greater pain intensity.
  Based on the distribution of pain VAS scores in post- surgical patients who described their postoperative pain intensity as none, mild, moderate, or severe, the following cut points on the pain VAS have been recommended: no pain (0-4 mm), mild pain (5-44 mm), moderate pain (45-74 mm), and severe pain (75-100 mm).
Pitsburg sleep quality index PSQI | 3 weeks
  it contains 19 self-rated questions and 5 self-rated by roommate (if available). The 19 self-rated questions are combined to 7 component scores each of which has 0-3 points. In all cases, a score of 0 indicates no difficulty while a score of 3 indicates severe difficulty. The seven score is then added to form one global score with a range of 0-21, 0 meaning no difficulty while 21 indicates severe difficulties in all areas

CONTACTS AND LOCATIONS:
Overall Officials: KINZA ANWAR, MS-OMPT, Principal Investigator — RIPHAH INTERNATIONAL UNIVERSITY,ISLAMABAD,PAKISTAN
Locations (1):
- Northwest Institute of Health Sciences and Northwest General Hospital Peshawar., Peshawar, Pakistan

IPD SHARING:
Plan to Share IPD: No